CLINICAL TRIAL: NCT04802044
Title: COVID-19, Aging, and Cardiometabolic Risk Factors (CARAMEL) Study: Integrating Aging, Cardiovascular, Metabolic, and Immunological Studies to Unravel COVID-19 Pathophysiology
Brief Title: COVID-19, Aging, and Cardiometabolic Risk Factors Study
Acronym: CARAMEL
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Indonesia University (Other)
Collaborators: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Dicky L. Tahapary, Principal Investigator, Indonesia University
Other Study IDs: CARAMEL
Record Dates: First submitted 2021-01-30; First posted 2021-03-17 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Covid19; Obesity; Diabetes Mellitus; Aging; Cardiometabolic Syndrome; Immune System Disorder
Keywords: COVID-19; adiposity; diabetes; insulin resistance; aging; inflammation; immune system
MeSH Terms: conditions — COVID-19; Obesity; Diabetes Mellitus; Metabolic Syndrome; Immune System Diseases; Insulin Resistance; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum Urine PBMC Nasal scrape Nasal swab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
COVID-19 pandemic has made a tremendous impact on Indonesian economic and health care system especially with the double burden of diseases facing by Indonesia as a developing country. The prevalence of non-communicable diseases such as obesity, type diabetes, and cardiovascular diseases is increasing. These diseases along with older age have been known as an established risk factors for higher mortality and severe clinical disease entity in COVID-19 infection. Although, there is still some part of patients with these co-morbidities that only present with mild symptoms when infected with SARS-CoV-2, even for some without any symptoms. Thus, it would be very interesting to evaluate how are these role of aging and cardiometabolic parameters in the clinical disease course of COVID-19 infection, and how are the relationship with the immune system.

DETAILED DESCRIPTION:
Indonesia is a country in transition where the burden of non-communicable diseases is taking over the infectious diseases problem, mostly due to the changes in lifestyle and increase in life expectancy.

However, the unprecedented rising numbers of COVID-19 patients in Indonesia has impacted the Indonesian healthcare system heavily. It has been reported that older age and the presence of cardiometabolic risk factors pose a poor prognostic factor of COVID-19. It is also important to note that in Indonesia, the presence of cardiometabolic risk factors is often observed at a younger age. Thus, this might also contribute to the higher mortality of COVID19 infected patients despite their relatively younger age in comparison to other countries. Nevertheless, specific data on the impact of aging and cardiometabolic risk factors on COVID-19 are fragmentary, justifying the achievement of a dedicated prospective observational study.

The CARAMEL study aims to specifically describe the phenotypic aging and cardiometabolic characteristics of patients with COVID-19 infection, in relation with the changes in the mucosal and systemic immune system. Particular attention will be devoted to obesity, central obesity, prediabetes, diabetes, hypertension, dyslipidemia, as well as anti-diabetic, antihypertensive, and anti-dyslipidemia therapies.

This study will provide answers to researchers, medical professionals, and especially patients, regarding the impact of aging and cardiometabolic risk factors for COVID-19 prognosis. This pilot study will be used for the development of new studies and for the establishment of recommendations for the care of patients with cardiometabolic risk factors and COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Patients newly diagnosed with COVID-19 at hospital setting or community screening, confirmed with biological proof (RT-PCR)

Exclusion Criteria:

* Subjects opposed to the use of their data
* Minors, adults under guardianship, protected persons
* History of malignancy
* History of autoimmune disease
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: COVID-19 patients in hospital and community setting
Sampling Method: Non-Probability Sample
Enrollment: 440 (Actual)
Dates: Start 2020-12-08 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Correlation of Body Mass Index with Clinical Disease Severity | Baseline
  To compare the body mass index, which calculated from body height (in meters) and body weight (in kilograms), in groups of COVID-19 patients with various disease severity based on WHO criteria
Correlation of Visceral Fat with Clinical Disease Severity | Baseline
  To compare the visceral fat that measures using a bio-impedance analyzer, in groups of COVID-19 patients with various disease severity based on WHO criteria
Correlation of Blood Glucose Levels with Clinical Disease Severity | Baseline
  To compare the random blood glucose levels during admission in groups of COVID-19 patients with various disease severity based on WHO criteria
Correlation of HbA1c with Clinical Disease Severity | Baseline
  To compare the HbA1c levels during admission in groups of COVID-19 patients with various disease severity based on WHO criteria

SECONDARY OUTCOMES:
Changes of Insulin Resistance Levels in COVID-19 Patients Overtime | Baseline, 6, and 12 month
  To compare the changes of HOMA-IR, a surrogate marker for whole-body insulin resistance which calculated from fasting blood glucose (IU/mL) and fasting insulin (mg/dL), between COVID-19 patients and healthy control subjects
Changes of Leptin/Adiponectin Ratio in COVID-19 Patients Overtime | Baseline, 6, and 12 month
  To compare the changes of leptin/adiponectin ratio, which calculated from leptin levels (ng/mL) divided by adiponectin levels (mikrogram/dL), between COVID-19 patients and healthy control subjects
Systemic Immune Profiles in Diabetic COVID-19 Patients | Baseline
  To compare the systemic immune profiles using mass cytometry between diabetic/COVID-19, non-diabetic/COVID-19, and healthy control subjects
Nasal Mucosal Immune Profiles in Diabetic COVID-19 Patients | Baseline
  To compare the nasal-mucosal immune profiles using mass cytometry between diabetic/COVID-19, non-diabetic/COVID-19, and healthy control subjects
Aging Parameter (ACE-2 gene expression) in COVID-19 Patients | Baseline
  To compare the nasal epithelial ACE-2 gene expression in groups of COVID-19 patients with various disease severity based on WHO criteria
Aging Parameter (Telomere Length) in COVID-19 Patients | Baseline
  To compare the aging parameter using telomere length in groups of COVID-19 patients with various disease severity based on WHO criteria
Immune Cells Exhaustion in COVID-19 Patients | Baseline
  To compare the immune cells exhaustion marker (T-cell immunoglobulin mucin-3/TIM-3 expressions) in groups of COVID-19 patients with various disease severity based on WHO criteria
Changes of Pro-Inflammatory Cytokine (IL-6) in COVID-19 Patients | Baseline, 1, 3, and 6 months
  To compare the changes of pro-inflammatory cytokine (IL-6) levels overtime, measured from the supernatant of stimulated PBMC isolation in groups of patients with various clinical disease severity based on WHO criteria
Changes of Anti-Inflammatory Cytokine (IL-10) in COVID-19 Patients | Baseline, 1, 3, and 6 months
  To compare the changes of anti-inflammatory cytokine (IL-10) levels overtime, measured from the supernatant of stimulated PBMC isolation in groups of patients with various clinical disease severity based on WHO criteria
Antibody Kinetics in COVID-19 Patients | Baseline, 1, 3, and 6 months
  To compare the changes of antibody titers in groups of patients with various clinical disease severity based on WHO criteria
Proportion of Long COVID Syndrome | 3, 6, and 12 months
  Percentage of COVID-19 patients still present with symptoms compared to whole study subjects

CONTACTS AND LOCATIONS:
Overall Officials: Dicky L Tahapary, Principal Investigator — Indonesia University
Locations (2):
- Indonesia (2):
  - Dr. Cipto Mangunkusumo National General Hospital, Jakarta Pusat, DKI Jakarta
  - Metabolic Disorder, Cardiovascular, and Aging Research Cluster IMERI-FKUI, Research Tower, 5th Floor, Jakarta Pusat, DKI Jakarta

REFERENCES:
- [Background] Liu K, Chen Y, Lin R, Han K. Clinical features of COVID-19 in elderly patients: A comparison with young and middle-aged patients. J Infect. 2020 Jun;80(6):e14-e18. doi: 10.1016/j.jinf.2020.03.005. Epub 2020 Mar 27. PMID 32171866
- [Background] Iannelli A, Favre G, Frey S, Esnault V, Gugenheim J, Bouam S, Schiavo L, Tran A, Alifano M. Obesity and COVID-19: ACE 2, the Missing Tile. Obes Surg. 2020 Nov;30(11):4615-4617. doi: 10.1007/s11695-020-04734-7. No abstract available. PMID 32451913
- [Background] Apicella M, Campopiano MC, Mantuano M, Mazoni L, Coppelli A, Del Prato S. COVID-19 in people with diabetes: understanding the reasons for worse outcomes. Lancet Diabetes Endocrinol. 2020 Sep;8(9):782-792. doi: 10.1016/S2213-8587(20)30238-2. Epub 2020 Jul 17. PMID 32687793
- [Background] Wu H, Ballantyne CM. Metabolic Inflammation and Insulin Resistance in Obesity. Circ Res. 2020 May 22;126(11):1549-1564. doi: 10.1161/CIRCRESAHA.119.315896. Epub 2020 May 21. PMID 32437299
- [Background] Andersen CJ, Murphy KE, Fernandez ML. Impact of Obesity and Metabolic Syndrome on Immunity. Adv Nutr. 2016 Jan 15;7(1):66-75. doi: 10.3945/an.115.010207. Print 2016 Jan. PMID 26773015
- [Background] Exley MA, Hand L, O'Shea D, Lynch L. Interplay between the immune system and adipose tissue in obesity. J Endocrinol. 2014 Nov;223(2):R41-8. doi: 10.1530/JOE-13-0516. Epub 2014 Sep 16. PMID 25228503
- [Background] Agrawal M, Kern PA, Nikolajczyk BS. The Immune System in Obesity: Developing Paradigms Amidst Inconvenient Truths. Curr Diab Rep. 2017 Aug 15;17(10):87. doi: 10.1007/s11892-017-0917-9. PMID 28812211
- [Background] Gerriets VA, MacIver NJ. Role of T cells in malnutrition and obesity. Front Immunol. 2014 Aug 11;5:379. doi: 10.3389/fimmu.2014.00379. eCollection 2014. PMID 25157251
- [Background] Han JM, Levings MK. Immune regulation in obesity-associated adipose inflammation. J Immunol. 2013 Jul 15;191(2):527-32. doi: 10.4049/jimmunol.1301035. PMID 23825387
- [Background] Rebello CJ, Kirwan JP, Greenway FL. Obesity, the most common comorbidity in SARS-CoV-2: is leptin the link? Int J Obes (Lond). 2020 Sep;44(9):1810-1817. doi: 10.1038/s41366-020-0640-5. Epub 2020 Jul 9. PMID 32647360
- [Background] Misumi I, Starmer J, Uchimura T, Beck MA, Magnuson T, Whitmire JK. Obesity Expands a Distinct Population of T Cells in Adipose Tissue and Increases Vulnerability to Infection. Cell Rep. 2019 Apr 9;27(2):514-524.e5. doi: 10.1016/j.celrep.2019.03.030. PMID 30970254
- [Background] Kwaifa IK, Bahari H, Yong YK, Noor SM. Endothelial Dysfunction in Obesity-Induced Inflammation: Molecular Mechanisms and Clinical Implications. Biomolecules. 2020 Feb 13;10(2):291. doi: 10.3390/biom10020291. PMID 32069832
- [Background] Li M, Qian M, Xu J. Vascular Endothelial Regulation of Obesity-Associated Insulin Resistance. Front Cardiovasc Med. 2017 Aug 9;4:51. doi: 10.3389/fcvm.2017.00051. eCollection 2017. PMID 28848738
- [Background] Engin A. Endothelial Dysfunction in Obesity. Adv Exp Med Biol. 2017;960:345-379. doi: 10.1007/978-3-319-48382-5_15. PMID 28585207
- [Background] Meyers MR, Gokce N. Endothelial dysfunction in obesity: etiological role in atherosclerosis. Curr Opin Endocrinol Diabetes Obes. 2007 Oct;14(5):365-9. doi: 10.1097/MED.0b013e3282be90a8. PMID 17940464
- [Background] van Deursen JM. The role of senescent cells in ageing. Nature. 2014 May 22;509(7501):439-46. doi: 10.1038/nature13193. PMID 24848057
- [Background] Ni W, Yang X, Yang D, Bao J, Li R, Xiao Y, Hou C, Wang H, Liu J, Yang D, Xu Y, Cao Z, Gao Z. Role of angiotensin-converting enzyme 2 (ACE2) in COVID-19. Crit Care. 2020 Jul 13;24(1):422. doi: 10.1186/s13054-020-03120-0. PMID 32660650
- [Background] Sungnak W, Huang N, Becavin C, Berg M, Queen R, Litvinukova M, Talavera-Lopez C, Maatz H, Reichart D, Sampaziotis F, Worlock KB, Yoshida M, Barnes JL; HCA Lung Biological Network. SARS-CoV-2 entry factors are highly expressed in nasal epithelial cells together with innate immune genes. Nat Med. 2020 May;26(5):681-687. doi: 10.1038/s41591-020-0868-6. Epub 2020 Apr 23. PMID 32327758
- [Background] Khemais-Benkhiat S, Idris-Khodja N, Ribeiro TP, Silva GC, Abbas M, Kheloufi M, Lee JO, Toti F, Auger C, Schini-Kerth VB. The Redox-sensitive Induction of the Local Angiotensin System Promotes Both Premature and Replicative Endothelial Senescence: Preventive Effect of a Standardized Crataegus Extract. J Gerontol A Biol Sci Med Sci. 2016 Dec;71(12):1581-1590. doi: 10.1093/gerona/glv213. Epub 2015 Dec 15. PMID 26672612
- [Background] Song J, Hu B, Qu H, Wang L, Huang X, Li M, Zhang M. Upregulation of angiotensin converting enzyme 2 by shear stress reduced inflammation and proliferation in vascular endothelial cells. Biochem Biophys Res Commun. 2020 May 7;525(3):812-818. doi: 10.1016/j.bbrc.2020.02.151. Epub 2020 Mar 10. PMID 32169277
- [Background] Bunyavanich S, Do A, Vicencio A. Nasal Gene Expression of Angiotensin-Converting Enzyme 2 in Children and Adults. JAMA. 2020 Jun 16;323(23):2427-2429. doi: 10.1001/jama.2020.8707. PMID 32432657
- [Background] Alsufyani HA, Docherty JR. The renin angiotensin aldosterone system and COVID-19. Saudi Pharm J. 2020 Aug;28(8):977-984. doi: 10.1016/j.jsps.2020.06.019. Epub 2020 Jul 2. PMID 32788834
- [Background] Al-Benna S. Association of high level gene expression of ACE2 in adipose tissue with mortality of COVID-19 infection in obese patients. Obes Med. 2020 Sep;19:100283. doi: 10.1016/j.obmed.2020.100283. Epub 2020 Jul 18. PMID 32835126
- [Background] Michalakis K, Ilias I. SARS-CoV-2 infection and obesity: Common inflammatory and metabolic aspects. Diabetes Metab Syndr. 2020 Jul-Aug;14(4):469-471. doi: 10.1016/j.dsx.2020.04.033. Epub 2020 Apr 29. PMID 32387864
- [Background] Telles S, Reddy SK, Nagendra HR. Obesity, Inflammation and Endothelial Dysfunction. J Chem Inf Model. 2019;53(9):1689-99.
- [Background] Cervia C, Nilsson J, Zurbuchen Y, Valaperti A, Schreiner J, Wolfensberger A, Raeber ME, Adamo S, Weigang S, Emmenegger M, Hasler S, Bosshard PP, De Cecco E, Bachli E, Rudiger A, Stussi-Helbling M, Huber LC, Zinkernagel AS, Schaer DJ, Aguzzi A, Kochs G, Held U, Probst-Muller E, Rampini SK, Boyman O. Systemic and mucosal antibody responses specific to SARS-CoV-2 during mild versus severe COVID-19. J Allergy Clin Immunol. 2021 Feb;147(2):545-557.e9. doi: 10.1016/j.jaci.2020.10.040. Epub 2020 Nov 20. PMID 33221383
- [Background] Peron JPS, Nakaya H. Susceptibility of the Elderly to SARS-CoV-2 Infection: ACE-2 Overexpression, Shedding, and Antibody-dependent Enhancement (ADE). Clinics (Sao Paulo). 2020;75:e1912. doi: 10.6061/clinics/2020/e1912. Epub 2020 May 15. PMID 32428113
- [Background] Lopes-Paciencia S, Saint-Germain E, Rowell MC, Ruiz AF, Kalegari P, Ferbeyre G. The senescence-associated secretory phenotype and its regulation. Cytokine. 2019 May;117:15-22. doi: 10.1016/j.cyto.2019.01.013. Epub 2019 Feb 16. PMID 30776684
- [Background] Asghar M, Yman V, Homann MV, Sonden K, Hammar U, Hasselquist D, Farnert A. Cellular aging dynamics after acute malaria infection: A 12-month longitudinal study. Aging Cell. 2018 Feb;17(1):e12702. doi: 10.1111/acel.12702. Epub 2017 Nov 16. PMID 29143441
- [Background] Pathai S, Lawn SD, Gilbert CE, McGuinness D, McGlynn L, Weiss HA, Port J, Christ T, Barclay K, Wood R, Bekker LG, Shiels PG. Accelerated biological ageing in HIV-infected individuals in South Africa: a case-control study. AIDS. 2013 Sep 24;27(15):2375-84. doi: 10.1097/QAD.0b013e328363bf7f. PMID 23751258
- [Background] van de Berg PJ, Griffiths SJ, Yong SL, Macaulay R, Bemelman FJ, Jackson S, Henson SM, ten Berge IJ, Akbar AN, van Lier RA. Cytomegalovirus infection reduces telomere length of the circulating T cell pool. J Immunol. 2010 Apr 1;184(7):3417-23. doi: 10.4049/jimmunol.0903442. Epub 2010 Feb 22. PMID 20176738
- [Background] Robinson MW, McGuinness D, Swann R, Barclay S, Mills PR, Patel AH, McLauchlan J, Shiels PG. Non cell autonomous upregulation of CDKN2 transcription linked to progression of chronic hepatitis C disease. Aging Cell. 2013 Dec;12(6):1141-3. doi: 10.1111/acel.12125. Epub 2013 Aug 12. PMID 23931242